CLINICAL TRIAL: NCT04452084
Title: Randomised Prospective Phase 2 Trial in Multiple Brain Metastases Comparing Outcomes Between Hippocampal Avoidance Whole Brain Radiotherapy With or Without Simultaneous Integrated Boost
Brief Title: Phase 2 Trial in Multiple Brain Metastases Outcomes With HA-SIB-WBRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singhealth Duke-NUS Oncology Academic Clinical Programme (ONCO ACP) (Unknown); Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA-SIB-WBRT
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Brain Metastases
Keywords: Whole Brain Radiotherapy; Brain metastases; Cognitive outcomes
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Masking Description: Blinding is not feasible in this study and will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Radiation: HA-WBRT
- Experimental Procedure (Experimental)
  Interventions: Radiation: HA-SIB-WBRT

INTERVENTIONS:
Radiation: HA-WBRT — The accepted standard HA-WBRT doses in the control arm are 30Gy in 10 fractions.
  Arms: Control
Radiation: HA-SIB-WBRT — The doses selected for experimental HA-SIB-WBRT arm are 30Gy in 10 fractions to the whole brain with 40 to 45Gy in 10 fraction SIB doses to tumours.
  Arms: Experimental Procedure

SUMMARY:
Recently, the evidence supports hippocampal avoidance with whole brain radiotherapy (HA-WBRT) as the recommended treatment option in patients with good prognosis and multiple brain metastases as it gives better neurocognitive preservation compared to historical whole brain radiotherapy controls. There is however often poor tumour control with this technique due to the low doses given. Stereotactic Radiosurgery (SRS), a form of focused radiotherapy which is given to patients who have a limited number of brain metastases, gives a higher radiation dose to the metastases resulting in better target lesion control. With improvements in radiation technology, advanced dose-painting techniques now allow a simultaneous integrate boost (SIB) dose to lesions whilst minimising doses to the hippocampus to potentially improve brain tumour control and preserve cognitive outcomes (HA-SIB-WBRT).

The Investigators believe that the SIB in HA-SIB-WBRT (experimental) will result in better functional and survival outcomes compared to HA-WBRT (control). Patients who are fit, have multiple brain metastases (5-25 lesions) and reasonable life expectancy (>6 months) will be recruited from NCCS over 2 years. Patients will be followed up the over the following year with imaging, toxicity data, quality of life, activities of daily living and cognitive measurements at set time points. The results will be compared across the 2 arms.

Patients with brain metastases are living longer. Maintaining functional independence and brain metastases control is thus increasingly important. Improved radiotherapy treatment techniques could provide better control and survival outcomes whilst maintain QoL and functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* 21-80 years old patients with radiological confirmed brain metastases (5-25 lesions)
* Histologically proven malignancy of primary cancer
* ECOG performance status ≤ 2
* Maximum lesion or cavity size ≤ 5cm

  * For patients with large (≥ 3cm) lesions, a neurosurgical consult is recommended as the risk of cerebral oedema and hydrocephalus is higher with RT. A Ventricular-peritoneal shunt/ surgical excision may be required prior to planning of RT
  * If brain surgery or other invasive procedures are performed, the treatment can only begin at least 2-weeks post-procedure
* Life expectancy of at least 6 months
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential
* Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control throughout protocol treatment
* Not recommended or does not want Stereotactic Radiosurgery (SRS)
* Agrees to be randomised to either HA-WBRT or HA-SIB-WBRT

Exclusion Criteria:

* Prior whole brain radiotherapy

  o Prior SRS is not an exclusion. Details of treatment must be recorded.
* Concurrent systemic cytotoxic treatment.

  o If patient is on systemic treatment a treatment break of at least 7 days for immunotherapy or chemotherapy and 3 days for targeted therapy is required before and after radiotherapy.
* Leptomeningeal disease
* Extensive extracranial disease, not controlled by systemic treatment
* Severe, active co-morbidity, defined as follows:

  * Major medical or psychiatric illness, which in the investigator's opinion would interfere with the completion of therapy and follow up or with full understanding of the risks and potential complications of the therapy;
  * Unstable angina and/or uncontrolled congestive heart failure;
  * Myocardial infarction within the last 6 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; note that patients switched from IV antibiotics and currently on oral antibiotics whose infection is assessed to be adequately treated or controlled are eligible.
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration;
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
  * Dementia, ongoing psychotic episodes or moderate-severe depression (PHQ-9).
  * Recent stroke in the past 3 months
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception;
* ECOG performance status >2 despite a duration of high dose steroids
* Symptomatic brain metastases limiting ADLs
* Rapid brain progression
* Patients unable to give informed consent
* Total tumour planning target volume (PTV) >60cc
* Radiological evidence of hydrocephalus
* Contraindication to Gadolinium contrast-enhanced MRI brain
* Patients who are unable to meet expected follow-up schedule (e.g. non-resident patients)
* Patients with diagnoses of small cell carcinoma, lymphoma or primary brain tumour

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Target lesion progression | From time of randomisation to target lesion progression, up to 6 months after last day of radiotherapy.

SECONDARY OUTCOMES:
Time to symptomatic brain metastases | From time of randomisation to symptomatic brain progression, up to 12 months after last day of radiotherapy.
Incidences of treatment-emergent adverse events (AE) | From time of randomisation to 12 months after last day of radiotherapy.
  Identified and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria.
Overall Survival | From time of randomisation to death from any cause, up to 12 months after last day of radiotherapy.
Progression Free Survival | From time of randomisation to overall progression, up to 12 months after last day of radiotherapy.
Cognitive function | From time of randomisation to 12 months after last day of radiotherapy.
  Assessed using Hopkins Verbal Learning Test

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Chia, MB ChB BAO, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Chia BSH, Leong JY, Ong ALK, Lim C, Poon SH, Chua MLK, Chua KLM, Kusumawidjaja G, Chua ET, Wong FY, Lee TS. Randomised prospective phase II trial in multiple brain metastases comparing outcomes between hippocampal avoidance whole brain radiotherapy with or without simultaneous integrated boost: HA-SIB-WBRT study protocol. BMC Cancer. 2020 Oct 30;20(1):1045. doi: 10.1186/s12885-020-07565-y. PMID 33126867